CLINICAL TRIAL: NCT03142386
Title: Pain and Quality of Life Management in Oncology Geriatric Patients With Osteopathic Manipulative Treatment: a Pilot Study
Brief Title: Osteopathic Manipulative Treatment in Oncology Patients' Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Chiara Arienti, PhD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Oncology and Osteopathy
Record Dates: First submitted 2017-04-28; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Geriatric Oncology; Osteopathy in Other Diseases Classified Elsewhere
Keywords: geriatric oncology; pain; osteopathic manipulative treatment; quality of life
MeSH Terms: conditions — Pain | interventions — Manipulation, Osteopathic; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT group (Experimental): Osteopathic manipulative treatment
  Interventions: Other: Osteopathic manipulative treatment
- Control Group (Active Comparator): Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Osteopathic manipulative treatment
  Arms: OMT group
Other: Physiotherapy
  Arms: Control Group

SUMMARY:
The aim of present study was to study the osteopathic manipulative effects on pain relief and quality of life improvement on hospitalized oncology geriatric patients. A non-randomized comparison trial was performed in Unit of Oncology Rehabilitation, Palazzolo Institute, Don Carlo Gnocchi Foundation ONLUS, Milan, Italy, from September 2015 to March 2016. 23 older oncology patients were unrolled and allocated in two experimental groups: study group (OMT group, N=12) underwent to osteopathic manipulative treatment associated to physiotherapy and control group (PT group, N = 11) underwent only physiotherapy. At enrollment (T0), 23 recruited oncology patients completed the socio-demographic forms and were evaluated, from external examiner, pain intensity and quality of life. All patients were revaluated at the end of treatment (T4) for quality of life and every week (T1, T2, T3 and T4) for pain intensity. Standard level of significance was p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* oncology patients
* male and female
* age≥65 years
* with a clinical prognosis of 6-24 months
* diagnosis of multifactorial hyperkinetic syndrome (i.e. metastatic surgery)
* pain intensity score higher than 3, measured with Numeric Rating Scale (NRS)

Exclusion Criteria:

* patients were receiving chemotherapy or radiotherapy treatment at the time of the study
* with mental disorders (MMSE<10)
* the presence of infection
* anticoagulation therapy
* cardiopulmonary disease
* clinical instability post-surgery.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pain | Once a week for a total 4 weeks
  Numeric Rating Scale (NRS) is a validated scale to measure the intensity of pain, with numbers between 0 and 10, with 0 representing absence of pain and 10 the worst possible pain experienced by the patient.

SECONDARY OUTCOMES:
Quality of life | At baseline and up to 4 weeks.
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQC30) is a validated multidimensional health-related quality of life (HRQOL) questionnaire composed of six functional scales, three symptom scales, and several additional single item scales.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Arienti, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arienti C, Bosisio T, Ratti S, Miglioli R, Negrini S. Osteopathic Manipulative Treatment Effect on Pain Relief and Quality of Life in Oncology Geriatric Patients: A Nonrandomized Controlled Clinical Trial. Integr Cancer Ther. 2018 Dec;17(4):1163-1171. doi: 10.1177/1534735418796954. Epub 2018 Aug 31. PMID 30168356